CLINICAL TRIAL: NCT04209257
Title: Functional Electrical Stimulation to Improve Crouch Gait in Cerebral Palsy
Brief Title: FES to Improve Crouch Gait in CP
Acronym: CP FES Walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Samuel C.K. Lee, PhD, PT, Principal Investigator, University of Delaware
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 71011-PHI
Record Dates: First submitted 2019-12-12; First posted 2019-12-24 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Cerebral Palsy; Gait
Keywords: Cerebral Palsy; Functional electrical stimulation; Neurotherapeutic
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Functional Electrical Stimulation protocol (Experimental): Participants will be evaluated with and without the use of functional electrical stimulation while walking to determine the neuroprosthetic and neurotherapeutic effects.
  Interventions: Device: Functional Electrical Stimulation.

INTERVENTIONS:
Device: Functional Electrical Stimulation. — Functional electrical stimulation - electrical stimulation applied to a muscle during an activity (i.e. ankle dorsiflexors during swing phase of gait). It assists / elicits muscle activation in order to achieve a task.

SUMMARY:
The overall goal of the proposed work is to develop and to assess the feasibility of using functional electrical stimulation (FES) system to improve crouch gait in individuals with cerebral palsy that may prevent the typical downward spiral of walking function decline in individuals with CP that occurs from adolescence into adulthood.

DETAILED DESCRIPTION:
Aim 1: To assess the feasibility of using a multiple channel FES system to produce an immediate neuroprosthetic effect to reduce crouch gait in children and adolescents with spastic diplegic CP.

Aim 2: To assess the feasibility of using a multiple channel FES system as a therapeutic training tool to produce lasting neurotherapeutic effects of diminished crouch gait in children and adolescents with CP.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-18
* Spastic CP (di-, tetra-, or triplegia)
* Levels I-II GMFCS classification
* Sufficient covering of the femoral head in the acetabulum (migration % < 40)
* Mild crouch gait (minimum knee flexion 21-40o during stance)
* Potential to gain > 20 degrees knee extension improvement in stance phase
* Minimum of 0o ankle dorsiflexion passive range of motion (PROM)
* Visual, perceptual, cognitive, and communication skills to follow multiple step commands for attending to exercise and data collection
* Seizure-free or well controlled seizures

Exclusion Criteria:

* Athetoid, ataxic, or hemiplegic CP
* Significant scoliosis (primary curve > 40°)
* Spinal fusions extending into the pelvis
* Severe tactile hypersensitivity
* Joint instability or dislocation in lower extremity
* Lower extremity surgery or fractures in the past year
* Botox injections to Lower extremity in the past 6 months
* Implanted medical device contraindicated with application of FES
* Severe spasticity in Lower extremity (Mod Ashworth 4)
* Lower extremity joint pain during walking
* Hx of pulmonary disease limiting exercise tolerance or Hx of cardiac disease
* Severely limited range of motion / contractures (>15o knee flex or >15o hip flex contractures)
* Pregnancy

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2012-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in the Muscle Tone | Change from the baseline Modified Ashworth Scale at 14 weeks (post training)
  We use the Modified Ashworth Scale to measure resistance to passive movement about a joint with varying degree of velocity (Muscle tone/spasticity). Score ranges from 0-4, with 6 choices where score of 0 means no increase in tone and score of 4 means rigid limb with no flexion or extension. Our training approach using repetitive electrical stimulation may also lower spasticity, which can also facilitate improved functional mobility.
Change in the Muscle Tone | Change from the baseline Modified Ashworth Scale at 27 weeks (Follow up)
  We use the Modified Ashworth Scale to measure resistance to passive movement about a joint with varying degree of velocity (Muscle tone/spasticity). Score ranges from 0-4, with 6 choices where score of 0 means no increase in tone and score of 4 means rigid limb with no flexion or extension. Our training approach using repetitive electrical stimulation may also lower spasticity, which can also facilitate improved functional mobility.
Metabolic Cost of Walking | Change from the baseline Metabolic Cost of Walking at 14 weeks (post training)
  Walking Energy Expenditure will be measured via indirect calorimetry at the subject's self-selected walking speed. The subject will walk on the treadmill while breathing into a VMax gas-dilution SensorMedics metabolic measurement system. The subject will warm up at a slow walking speed for 3 minutes, walk for approximately 5 minutes at the subject's self-selected walking speed until steady state is reached, and then sit for a 3-minute cool down. The metabolic cost of walking is computed over the 5-minute walking period.
Metabolic Cost of Walking | Change from the baseline Metabolic Cost of Walking at 27 weeks (Follow up)
  Walking Energy Expenditure will be measured via indirect calorimetry at the subject's self-selected walking speed. The subject will walk on the treadmill while breathing into a VMax gas-dilution SensorMedics metabolic measurement system. The subject will warm up at a slow walking speed for 3 minutes, walk for approximately 5 minutes at the subject's self-selected walking speed until steady state is reached, and then sit for a 3-minute cool down. The metabolic cost of walking is computed over the 5-minute walking period.
Change in the Walking Speed | Change from the baseline Walking speed at 14 weeks (Post training)
  Walking Speed is measured via the 10-meter walk test. This time taken to complete the task is used to compute the average walking speed referred to as "self-selected" walking speed.
Change in the Walking Speed | Change from the baseline Walking speed at 27 weeks (Follow up)
  Walking Speed is measured via the 10-meter walk test. This time taken to complete the task is used to compute the average walking speed referred to as "self-selected" walking speed.
Change in the Walking Distance | Change from the baseline Walking Distance at 14 weeks (Post training)
  Walking distance (in a fixed period of time) is an indicator of endurance. Walking Distance is measured via the 6-minute walk test. Improved motor learning and gait biomechanics from the training methods would improve gait efficiency and thus, endurance.
Change in the Walking Distance | Change from the baseline Walking Distance at 27 weeks (Follow up)
  Walking distance (in a fixed period of time) is an indicator of endurance. Walking Distance is measured via the 6-minute walk test. Improved motor learning and gait biomechanics from the training methods would improve gait efficiency and thus, endurance.
Change in Gross Motor Function Measure | Change from the baseline GMFM score at 14 weeks (Post training)
  Gross Motor Function will be assessed via sections D and E of the Gross Motor Function Measure (GMFM) test. This test is designed to evaluate changes in gross motor function over time of children with CP.
Change in Gross Motor Function Measure | Change from the baseline GMFM score at 27 weeks (Follow up)
  Gross Motor Function will be assessed via sections D and E of the Gross Motor Function Measure (GMFM) test. This test is designed to evaluate changes in gross motor function over time of children with CP.
Change in the Timed Up-And-Go (TUG time) | Change from the baseline Time Up and Go time at 14 weeks (Post training)
  Timed Up-And-Go (TUG) is a measure designed to assess functional mobility and balance. The subjects will be seated on an adjustable bench such that the knees and angles are at 90 degrees. Subjects will be timed as they rise, walk 3 meters, turn around, return to the bench and sit down again.assessing the impact of anticipated improvements in motor control and gait biomechanics.
Change in the Timed Up-And-Go (TUG time) | Change from the baseline Time Up and Go time at 27 weeks (Follow up)
  Timed Up-And-Go (TUG) is a measure designed to assess functional mobility and balance. The subjects will be seated on an adjustable bench such that the knees and angles are at 90 degrees. Subjects will be timed as they rise, walk 3 meters, turn around, return to the bench and sit down again.assessing the impact of anticipated improvements in motor control and gait biomechanics.
Change in the Mini Balance Evaluation Systems Test Score | Change from the baseline Mini BESTest score at 14 weeks (Post training)
  Balance Evaluation Systems Test (BESTest) is a measure of balance function. The BESTest will allow for assessing the impact of anticipated improvements in motor control and gait biomechanics from training on balance. The test has a maximum score of 28 points and minimum score of zero. Score of 28 means highest level of function and 0 means lowest level of function.
Change in the Mini Balance Evaluation Systems Test Score | Change from the baseline Mini BESTest score at 27 weeks (Follow up)
  Balance Evaluation Systems Test (BESTest) is a measure of balance function. The BESTest will allow for assessing the impact of anticipated improvements in motor control and gait biomechanics from training on balance. The test has a maximum score of 28 points and minimum score of zero. Score of 28 means highest level of function and 0 means lowest level of function.
Change in the Electromyography | Change from the baseline Muscle activation at 14 weeks (Post training)
  Muscle activation timing measured with Electromyography during gait analysis allows for mechanistic study of anticipated improvements in motor control and gait as well as comparison to typical norms.
Change in the Electromyography | Change from the baseline Muscle activation at 27 weeks (Follow up)
  Muscle activation timing measured with Electromyography during gait analysis allows for mechanistic study of anticipated improvements in motor control and gait as well as comparison to typical norms.
Changes in the Activities-Specific Balance Scale Score | Change from the baseline ABC scale score at 14 weeks (Post training)
  The Activities-Specific Balance Scale (ABC Scale) survey allows measurement of perceived functional mobility by assessing balance confidence to perform daily activities of living without falling. 16 items are rated on a rating scale with range of 0-100. Score of 0 means no confidence and 100 means complete confidence. Average score of 16 items is the overall score. Such measures will assess the impact of anticipated improvements in motor control and gait bio-mechanics from training.
Changes in the Activities-Specific Balance Scale Score | Change from the baseline ABC scale score at 27 weeks (Follow up)
  The Activities-Specific Balance Scale (ABC Scale) survey allows measurement of perceived functional mobility by assessing balance confidence to perform daily activities of living without falling. 16 items are rated on a rating scale with range of 0-100. Score of 0 means no confidence and 100 means complete confidence. Average score of 16 items is the overall score. Such measures will assess the impact of anticipated improvements in motor control and gait bio-mechanics from training.
Changes in the Participation in Life Events survey score | Change from the baseline LIFE-H scale score at 14 weeks (Post training)
  Participation in life events (LIFE-H) survey measures how much a person is engaging or participating with their peers and community. Weighted score ranges between 0-10 with 0 score being no accomplishment and 10 means complete accomplishment. Such measures will assess the impact of anticipated improvements in motor control and gait biomechanics from training.
Changes in the Participation in Life Events survey score | Change from the baseline LIFE-H scale score at 27 weeks (Follow up)
  Participation in life events (LIFE-H) survey measures how much a person is engaging or participating with their peers and community. Weighted score ranges between 0-10 with 0 score being no accomplishment and 10 means complete accomplishment. Such measures will assess the impact of anticipated improvements in motor control and gait biomechanics from training.
Change in Piers-Harris Children's Self-Concept Scale score | Change from the baseline Piers-Harris Children's Self-Concept scale score at 14 weeks (Post training)
  Self-Perception will be measured via the Piers-Harris Children's Self-Concept Scale, Second Edition (Piers-Harris 2). This test is designed to measure self-concept as reported by the individual. It measures physical and emotional well-being and self-esteem and will allow assessment of the impact of anticipated improvements in motor control and gait biomechanics from training. The tool consists of 60 items that require the respondent to respond by circling "Yes" or "No." Raw scores are converted to standardized t-scores (mean = 50, standard deviation = 10) and percentile ranks. T-Score ranges for the total scale are: <29T is very low, 30T-39T is low, 40T-44T is low average, 45T-55T average, 56T-59T- is high average, 60T-69T is high and > 70T is very high. For the six subscales T-Score ranges < 29T is very low, 30T-39T is low, 40T-44T is low average, 45T-55T is average and > 56T is above average.
Change in Piers-Harris Children's Self-Concept Scale score | Change from the baseline Piers-Harris Children's Self-Concept scale score at 27 weeks (Follow up)
  Self-Perception will be measured via the Piers-Harris Children's Self-Concept Scale, Second Edition (Piers-Harris 2). This test is designed to measure self-concept as reported by the individual. It measures physical and emotional well-being and self-esteem and will allow assessment of the impact of anticipated improvements in motor control and gait biomechanics from training. The tool consists of 60 items that require the respondent to respond by circling "Yes" or "No." Raw scores are converted to standardized t-scores (mean = 50, standard deviation = 10) and percentile ranks. T-Score ranges for the total scale are: <29T is very low, 30T-39T is low, 40T-44T is low average, 45T-55T average, 56T-59T- is high average, 60T-69T is high and > 70T is very high. For the six subscales T-Score ranges < 29T is very low, 30T-39T is low, 40T-44T is low average, 45T-55T is average and > 56T is above average.
Change in Joint angles | Change from the baseline Joint angles at 14 weeks (Post training)
  Hip, Knee and Ankle Joint Angles (Kinematic data) are measured using Instrumented gait analysis (Motion capture analysis system) during seven different gait phases.
Change in Joint angles | Change from the baseline joint angles at 27 weeks (Follow up)
  Hip, Knee and Ankle Joint Angles (Kinematic data) are measured using Instrumented gait analysis (Motion capture analysis system) during seven different gait phases.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Lee, PT, PhD, Principal Investigator — Shriners Hospital for Children & University of Delaware
Locations (1):
- Shriners Hospitals for Children, Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The proposed experiments will generate data for publications in high quality peer reviewed journals. We will also present our findings at national meetings of neurorehabilitation scientists and clinicians and neuroscience and motor control meetings. To have the most impact, it is important that we present our findings to both clinicians and scientists, therefore, in addition to these standard approaches, we will seek out regular opportunities to present both the rationale and results of our work to local and regional clinicians as well as local and regional stroke support groups.
  Once the primary hypotheses of the current proposal are tested, all data will be de-identified and be deposited in the DASH (The Data and Specimen Hub) repository.
Supporting Information: Study Protocol, CSR
Time Frame: Study protocol and data will be shared on publication of primary results

REFERENCES:
- See also: Dr. Lee's current research studies — http://sites.udel.edu/pt/dr-samuel-lee/